CLINICAL TRIAL: NCT03005821
Title: Chinese Pediatric Massage on Children With Acute Diarrhea: a Randomized Sham Massage Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Dongguan Kanghua Hospital (Other)
Responsible Party: Principal Investigator, Darong Wu, MD, PhD, Director,Program for Outcome Assessment in TCM, Professor, Chief Physician, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013B032500014
Record Dates: First submitted 2016-12-25; First posted 2016-12-29 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Diarrhea
Keywords: pediatric massage; Tuina therapy; acute diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pediatric massage (Experimental): Patients will receive Montmorillonite Powder and racecadotril granules as usual care according to different age or weight. Intravenous infusion, Oral Rehydration Salts (ORS), Zn,and antibiotics will be used if the pediatrician in charge considers necessary. Patients will receive Chinese pediatric massage once per day and for three days continuously. A cloak which can cover the child's hands and upper body will be required to put on, all the manipulations will be done under the cloak. Six acupoints will be adopted,i.e. Neibagua, Dachang,Xiaochang, Banmen, Fu, Tuishang Qijiegu. Each visit, children who are under 2 years old will receive manipulations on Neibagua for 500 times, 300 times for the other 5 acupoints each; if they are from 2-3 years old, the manipulations on Neibagua will be 700 times and 500 times for the other 5 acupoints respectively; while the manipulations on Neibagua will be 1000 times, and 800 times for the other 5 acupoints if the children are from 4-6 years old.
  Interventions: Other: Chinese pediatric massage therapy + usual care
- sham massage (Sham Comparator): Patients will receive the same usual care as the experimental group. For the sham massage, the therapist will use one hand to hold the childrens' hand or just put one hand on childrens' body and the other hand will do the manipulations on the therapist's own hand instead childrens' hand or childrens' body. Patients will be required to put on the same kind of cloak as that for the the experimental group, all the manipulations will be done under the cloak. The manipulation times for each acupoints will be the same as those for experimental group in accordance with different age. The sham massage will be given once per day for 3 days continuously.
  Interventions: Other: Sham massage therapy + usual care

INTERVENTIONS:
Other: Chinese pediatric massage therapy + usual care
  Arms: pediatric massage
Other: Sham massage therapy + usual care
  Arms: sham massage

SUMMARY:
The purpose of this study is to evaluate the efficacy of Chinese pediatric massage as an add-on therapy while comparing with sham massage both on the basis of usual care for 0-6 years old children with acute diarrhea.

DETAILED DESCRIPTION:
Chinese pediatric massage has been practised as an option for the treatment of pediatric diarrhea for hundreds of years (since Ming Dynasty). The history of Chinese pediatric massage for health promotion is much longer, it can be traced back to more than one thousand years ago (652 AD). Many of the acupoints adopted in Chinese pediatric massage are unique if it is compared with those for adult massage. The manipulation is found to be easily accepted by children, as the strength of massage is gentle and soft. No severe adverse reaction in regards of Chinese pediatric massage was reported, the mild adverse reaction such as skin abrasion can be completely avoided with correct operating instructions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's symptoms meet the diagnosis criteria of acute diarrhea.
2. The occurrence of diarrhea is no more than 72 hours.
3. Stool frequency is equal or more than 5 times a day.
4. Subject has not been involved in any other clinical trials at the same period of time.
5. Subject's guardian may coordinate during the clinical trial.
6. Subject's guardian have signed the informed consent.

Exclusion Criteria:

1. A history of experiencing Chinese pediatric massage on hands
2. Subject has cholera or malaria
3. Subject with the following conditions on the manipulating part: phlebitis，open wound，fracture，tissue damage
4. Subject has the follow complications: severe dehydration，metabolic acidosis，disorders of consciousness, seizures or twitching, shock, azotemia

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2017-01; Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Diarrhea days | Within 14 days, the period of days from baseline to the first day that the diarrhea time reduces to equal to or less than 2 times per day.
The diarrhea times | On the 3rd day.
  The baseline and the 1st day of intervention are on the same day.

SECONDARY OUTCOMES:
Global change rating | On the 7th day and 14th day from baseline (the baseline and the 1st day of intervention are on the same day).
  much better，slightly better，unchanged，slightly worse，much worse
Period of days when the stool character turns to normal | Within 14 days, the period of days from baseline to the first day that the stool character turns to normal.
Incidence of Treatment-Emergent Adverse Events | Within 14 days
  monitor adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguan Kanghua Hospital, Dongguan, Guangdong, China

REFERENCES:
- [Derived] Lu T, Yin L, Chen R, Zhang H, Cai J, Li M, Dai L, Zhu C, Zhang Y, Xiang F, Wang L, Li L, Wang L, Wu D. Chinese pediatric Tuina on children with acute diarrhea: a randomized sham-controlled trial. Health Qual Life Outcomes. 2021 Jan 6;19(1):4. doi: 10.1186/s12955-020-01636-1. PMID 33407547
- [Derived] Lu T, Zhang H, Yin L, Cai J, Li M, Dai L, Zhu C, Zhang Y, Xiang F, Wang L, Li L, Wang L, Wu D. Chinese pediatric Tuina on children with acute diarrhea: study protocol for a randomized sham-controlled trial. Trials. 2019 Dec 9;20(1):689. doi: 10.1186/s13063-019-3818-1. PMID 31815655